CLINICAL TRIAL: NCT02477917
Title: A Multicenter, Open Clinical Trial With Subcutaneous Immunotherapy in Depot in Patients With Rhinoconjunctivitis Sensitized to Parietaria Judaica
Brief Title: A Multicenter, Open Trial With Subcutaneous Immunotherapy (SCIT) in Patients With Rhinoconjunctivitis Sensitized to Parietaria Judaica
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roxall Medicina España S.A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-PAR-DEPOT
Record Dates: First submitted 2015-06-01; First posted 2015-06-23 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Rhinoconjunctivitis
Keywords: allergy; SCIT
MeSH Terms: conditions — Hypersensitivity | interventions — Parietaria judaica pollen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allergovac depot (Experimental): Allergovac depot with Parietaria judaica pollen extract
  Interventions: Biological: Allergovac depot with Parietaria judaica pollen extract

INTERVENTIONS:
Biological: Allergovac depot with Parietaria judaica pollen extract — Subcutaneous immunotherapy in depot presentation in a rapid dose escalation scheme: 6 weekly dose increasing injections at the initiation phase plus 3 maintenance monthly injections

SUMMARY:
The study was designed according to the draft of allergenic product regulation published by Spanish Regulatory Agency. The aim of the study is to evaluate the safety and tolerability of subcutaneous immunotherapy with Parietaria judaica pollen extract in patients with rhinoconjunctivitis with or without associated mild asthma. In addition, surrogate efficacy parameters will be evaluated: immunoglobulin level changes and skin reactivity.

DETAILED DESCRIPTION:
Parietaria judaica is a weed widespread throughout the Mediterranean área. Prevalence of sensitization to Parietaria judaica's pollen is very high in the Mediterranean areas, reaching 41.4% among allergic patients on the Spanish Mediterranean coast.

The study has been designed as an open trial which will be conducted in 4 Spanish sites.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must sign the informed consent form.
2. Patients must be between 18 and 60 years of age.
3. Patients with seasonal allergic rhinoconjunctivitis against Parietaria judaica during a minimum of 2 years prior to study participation. Although allergic rhinoconjunctivitis is the pathology under study, the inclusion of patients with mild concomitant asthma is allowed (GINA 2013).
4. Patients who obtained a prick test result ≥ 3 mm diameter to Parietaria judacia. Positive and negative control of the test should give consistent results.
5. Patients with specific immunoglobulin E ≥ class 2 (CAP/PHADIA) to Parietaria judaica.
6. Patients sensitized to Parietaria judaica with clinically relevant symptoms in which treatment with Parietaria judaica 100% vaccine is indicated.
7. Women of childbearing potential must have a negative urine pregnancy test at Screening visit/Visit 0.
8. Women of childbearing potential must agree to use an appropriate contraception method during the study if they are sexually active.

Exclusion Criteria:

1. Patients who received immunotherapy in the previous 5 years for Parietaria judaica or fo rany allergen with cross reactivity or patients that are currently receiving immunotherapy for any allergen.
2. Patients with severe asthma or forzed expiratoy volumen in 1 second FEV1< 70% even if the are pharmacologically controlled .
3. Patients with: immunological, cardiac, renal or hepatic illnesses or any other medical condition that the investigator deems relevant so as to interfere with the study.
4. Patients with a previous history of anaphylaxis
5. Patients with chronic urticaria,
6. Patients with moderate to severe atopic dermatitis
7. Patients who have participated in another clinical trial within 3 month prior to enrolment.
8. Patients under treatment with tricyclic antidepressives, phenothiazines , β-blockers, or Angiotensin Converting Enzyme Inhibitors (ACEI)
9. Female patients who are pregnant or breast-feeding
10. Patient who does not attend the visits
11. Patient's lack of collaboration or refusal to participate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number and severity of adverse reactions as a measure of Safety and tolerability | across 17 weeks treatment period

SECONDARY OUTCOMES:
Immunoglobulin changes from baseline | At baseline and 1 week after last administered dose
Skin reactivity changes from baseline | At baseline and 1 week after last administered dose

CONTACTS AND LOCATIONS:
Overall Officials: Araitz Landeta, Study Chair — Roxall Medicina España S.A
Locations (4):
- Spain (4):
  - Hospital Vega Baja, Orihuela, Alicante
  - Hospital de Manises, Manises, Valencia
  - Hosptal de Sagunto, Sagunto, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia